CLINICAL TRIAL: NCT06730516
Title: Optic Nerve Head Perfusion Following Treatment with Latanoprost 0.005% Versus Brimionidin Tartrate 0.2% in Primary Open Angle Glaucoma: an Optical Coherence Tomography Angiography Study
Brief Title: Optic Nerve Perfusion Following Treatment with Latanoprost Versus Brimionidin Tartrate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #454/25-June-2024.; Zagazig University (Registry Identifier: Institutional review board of zagazig university)
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma
Keywords: Latanoprost; Brimonidine
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Intervention Model Description: This prospective interventional randomized study included 56 naive patients recently diagnosed with bilateral primary open angle glaucoma equally divided into two groups with 28 patients in each group. Nine patients, five in group (1) and four in group (2) were excluded due to poor quality OCTA images or non-compliance). Group (1) included 23 patients (46 eyes) treated with Latanoprost 0.005 % while 24 patients (48 eyes) received treatment with Brimonidin tartrate 0.2% in group (2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Latanoprost (Xalatan) (Experimental): Group (1) included 23 patients (46 eyes) treated with Latanoprost 0.005 %
  Interventions: Drug: Latanoprost (Xalatan)
- Brimonidine 0.2% (Experimental): 24 patients (48 eyes) received treatment with Brimonidin tartrate 0.2% in group (2)
  Interventions: Drug: Brimonidine 0.2 %

INTERVENTIONS:
Drug: Latanoprost (Xalatan) — latanoprost 0.005
  Arms: Latanoprost (Xalatan)
Drug: Brimonidine 0.2 % — Brimonidine0.2
  Arms: Brimonidine 0.2%

SUMMARY:
This study aimed to evaluate the effects of topical Latanoprost 0.005 % versus Brimionidin tartrate 0.2% on perfusion of optic nerve head This prospective interventional randomized study included 56 naive patients recently diagnosed with bilateral primary open angle glaucoma equally divided into two groups with 28 patients in each group

DETAILED DESCRIPTION:
This study aimed to evaluate the effects of topical Latanoprost 0.005 % versus Brimionidin tartrate 0.2% on perfusion of optic nerve head This prospective interventional randomized study included 56 naive patients recently diagnosed with bilateral POAG equally divided into two groups with 28 patients in each group. The whole VD was increased and also increased in all four nasal, temporal, superior, and inferior quadrants around optic disc from the initial vessel density before treatment (p<0.001) in both groups significantly with superior improvement in group (1) compared to group (2) that was statistically significant

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years newly diagnosed naive patients with POAG

Exclusion Criteria:

* optic nerve lesions other than glaucomatous changes patients with previous glaucoma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
OPTIC NERVE PERFUSION using OCT angiography numerical analysis system presented in % | 3 months
  perfusion of optic nerve head in patients with primary open angle glaucoma (POAG) using optical coherence tomography angiography (OCTA).

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine A Deiaeldin, MD, Study Director — Zagazig University; Hani elbialy, MD, Study Director — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No